CLINICAL TRIAL: NCT05904106
Title: Venetoclax Plus Azacitidine Versus Standard Intensive Chemotherapy for Patients With Newly Diagnosed Acute Myeloid Leukemia (AML) and NPM1 Mutations Eligible for Intensive Treatment
Brief Title: Venetoclax Plus Azacitidine Versus Intensive Chemotherapy for Fit Patients With Newly Diagnosed NPM1 Mutated AML
Acronym: VINCENT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: University Hospital Heidelberg (Other); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUD-VINC01-080
Record Dates: First submitted 2023-05-25; First posted 2023-06-15 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; NPM1; venetoclax; azacitidine; Measurable Residual Disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — venetoclax; Azacitidine; Gemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ven+Aza arm (Experimental): non-intensive treatment: venetoclax plus azacitidine
  Interventions: Drug: Venetoclax plus Azacitidine
- SOC arm (Active Comparator): standard of care treatment: intensive chemotherapy plus gemtuzumab ozogamicin
  Interventions: Drug: standard of care chemotherapy plus gemtuzumab ozogamicin

INTERVENTIONS:
Drug: Venetoclax plus Azacitidine — Induction cycle 1:
  100 mg venetoclax p.o. on day 1; 200 mg venetoclax p.o. on day 2; 400 mg venetoclax p.o. on days 3-28; 75 mg/m^2 azacitidine s.c. on days 1-7
  Induction cycles 2-3:
  400 mg venetoclax p.o. on days 1-28; 75 mg/m^2 azacitidine s.c. on days 1-7
  Postremission cycles 1-9:
  400 mg venetoclax p.o. on days 1-28; 75 mg/m^2 azacitidine s.c. on days 1-7
  Arms: Ven+Aza arm
Drug: standard of care chemotherapy plus gemtuzumab ozogamicin — Induction cycle 1:
  200 mg/m^2 cytarabine cont inf i.v. on days 1-7; 60 mg/m^2 daunorubicin i.v. on days 3-5; 3 mg/m^2 (max 1 vial) gemtuzumab ozogamicin i.v. on days 1+4+7
  Induction cycle 2 (patients not in remission, moderate or non-responders):
  3000/1000 mg/m^2 cytarabine i.v. BID on days 1-3; 10 mg/m^2 mitoxantrone i.v. on days 3-5
  Postremission cycles 1-3:
  3000/1000 mg/m^2 cytarabine i.v. BID on days 1-3
  Arms: SOC arm

SUMMARY:
This phase II clinical trial evaluates the efficacy and tolerability of the non-intensive treatment with venetoclax and the hypomethylating agent azacitidine as compared to the standard of care chemotherapy plus gemtuzumab ozogamicin in newly diagnosed NPM1 mutated AML patients fit for intensive chemotherapy.

DETAILED DESCRIPTION:
AML is a heterogeneous disease of malignant early myeloid cells with a poor prognosis. Currently the only potentially curative treatment for patients with AML is intensive induction chemotherapy with 7 days of standard-dose cytarabine plus 3 days of an anthracyclin (7+3) followed either by several courses of consolidation chemotherapy with high-dose cytarabine or by allogeneic stem cell transplantation as standard of care (SOC). Complete remission (CR) is achieved in 60-80% of younger patients (aged 16-60 years) and in around 50% of older patients aged ≥ 60 years by this induction chemotherapy. However, this induction chemotherapy is toxic, due to prolonged myelosuppression with resulting infectious complications and organ toxicity with severe nausea, mucositis, colitis and cardiotoxicity. Each cycle of this intensive chemotherapy usually results in prolonged hospitalization of the patients and requires extensive supportive care with blood products and anti-infective agents. In addition, patients treated with intensive induction chemotherapy are at increased risk for several serious long-term side effects including cardiac and neurological sequelae, infertility and secondary cancers. The high toxicity burden in general and cardiovascular toxicity specifically consistently increase total costs in intensive induction and consolidation chemotherapy. From this perspective there is a need for therapies with lower toxicity and better efficacy.

Due to the high risk of early mortality, older patients and those with severe pre-existing conditions are typically treated with non-intensive chemotherapy with either low-dose cytarabine (LDAC) or a hypomethylating agent (HMA) either azacitidine or decitabine.While these treatments offer at best modest efficacy with CR rates of only 10%-30% and median overall survival of 6-12 months, combinations with the B-cell lymphoma-2 inhibitor venetoclax have been shown to produce CR rates between 50-75% in patients not eligible for intensive chemotherapy. The best response of venetoclax-based regimens with response rates up to 93% and two-year overall survival of 75% has been found among others in the large group of AML patients with mutations in the NPM1 gene. Standard intensive treatment in NPM1 mutated AML patients without adverse risk features usually consisting of standard of care chemotherapy plus gemtuzumab ozogamicin (GO) induces CR rates around 85%, and leads to a 5-year overall survival of around 40% - 50%.The rate and durability of response to venetoclax-based combinations in single arm studies with NPM1 mutated AML patients compared favourably with outcomes from intensive chemotherapy. A retrospective analysis in elderly AML patients with NPM1 mutation found remission rates of 73% in the entire cohort and 96 % in patients > 65 years. The venetoclax-based combination with the HMA azacitidine is generally well tolerated and has a better safety profile than intensive chemotherapy.

Based on these available clinical data it is postulated that non-intensive treatment with venetoclax plus azacitidine in NPM1 mutated fit AML patients may be equivalent or superior to the standard intensive treatment in terms of remission rates, relapse-free survival, treatment related mortality and health-related quality of life. This randomised controlled phase II trial (VINCENT) is to evaluate the efficacy and tolerability of the non-intensive treatment with venetolcax and azacitidine (Ven+Aza arm) in a wide age-range of newly diagnosed NPM1 mutated AML patients fit for intensive chemotherapy in comparison to standard of care chemotherapy plus GO (SOC arm).

ELIGIBILITY:
Inclusion Criteria:

1. A signed informed consent
2. Newly diagnosed CD33-positive AML with NPM1 mutation according to WHO criteria
3. Age 18-70 years
4. Fit for intensive chemotherapy, defined by

   * ECOG performance status of 0-2
   * Adequate hepatic function: ALAT/ASAT/Bilirubin ≤ 2.5 x ULN unless considered due to leukemic organ involvement Note: Subjects with Gilbert's Syndrome may have a bilirubin > 2.5 × ULN per discussion between the investigator and Coordinating investigator.
   * Adequate renal function assessed by serum creatinine ≤ 1.5x ULN OR creatinine clearance (by Cockcroft Gault formula) ≥ 50 mL/min
5. WBC < 25 x 109/L (<25,000/µL), prior hydroxyurea is permitted to meet this criterion
6. Ability to understand and the willingness to sign a written informed consent.
7. Male subjects must agree to refrain from unprotected sex and sperm donation from time point of signing the informed consent until 7 months after the last dose of study drug.
8. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 72 hours before first dose of study drug.

Exclusion Criteria:

1. Activating FLT3 mutation
2. Relapsed or refractory AML
3. AML after antecedent myelodysplasia (MDS) with prior cytotoxic treatment
4. Prior history of malignancy, other than MDS, unless the subject has been free of the disease for ≥ 1 year prior to start of study treatment (exceptions are basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or of the breast, incidental histologic finding of prostate cancer (T1a or T1b using the tumor, node, metastasis clinical staging system))
5. Previous treatment with HMA or venetoclax
6. Previous treatment for AML except hydroxyurea
7. Cumulative previous exposure to anthracyclines of > 200 mg/m^2 doxorubicin equivalents
8. CNS involvement or extramedullary disease only
9. Known hypersensitivity to excipients of the preparation or any agent given in association with this study including venetoclax, azacitidine, cytarabine, daunorubicin, gemtuzumab-ozogamicin, or mitoxantrone
10. Known positivity for human immunodeficiency virus (HIV) and History of active or chronic infectious hepatitis unless serology demonstrates clearance of infection (i.e.

    PCR undetectable viral load for hepatitis).
11. Inability to swallow oral medications
12. Any malabsorption condition
13. Cardiovascular disability status of New York Heart Association (NYHA) Class ≥ 2; unstable coronary artery disease (MI more than 6 months prior to study entry is permitted); serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.

    Note: Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or anginal pain.
14. Chronic respiratory disease that requires continuous oxygen use
15. Substance abuse, medical, psychological, or social conditions that may interfere with the subject's cooperation with the requirements of the trial or evaluation of the study results
16. Simultaneous participation in another interventional clinical trial
17. Pregnant or breastfeeding women. Breastfeeding has to be discontinued before onset of and during treatment and should be discontinued for at least 3 months after end of treatment.
18. Patients who are unwilling to follow strictly highly effective contraception requirements including hormonal contraceptives with an Pearl Index < 1% per year in combination with a barrier method from time point of signing the informed consent until 7 months after the last dose of study drug unless one of the following criteria is met:

    * post-menopausal (12 months natural amenorrhea or 6 months amenorrhea with serum FSH > 40 U/ml)
    * postoperative (6 weeks after bilateral ovarectomy with or without hysterectomy)
    * medically confirmed ovarian failure
    * vasectomy Note: At present, it is not known whether the effectiveness of hormonal contraceptives is reduced by venetoclax. For this reason, women must use a barrier method in addition to hormonal contraceptive methods.
19. History of clinically significant liver cirrhosis (e.g., Child-Pugh class B and C)
20. Live-virus vaccines given within 28 days prior to the initiation of study treatment Note: corona vaccines are not live-virus vaccines and are excluded from this criterion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-04-07 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
modified event-free survival (mEFS) | time interval from date of randomization until either primary treatment failure or hematologic relapse or molecular failure or death, whichever occurs first
  * Failure to achieve a CR/CRi/CRh after a maximum of two induction cycles in the control arm (SOC) or three induction cycles in the investigational arm (VEN+AZA), i.e. primary induction failure
  * Hematologic relapse after previous CR/CRi/CRh
  * Molecular failure, defined as either
    * Molecular progression, defined as confirmed ≥ 1 log10 increase of NPM1 MRD level in any two samples in a patient without prior MRD negativity or
    * Molecular relapse after previous MRD negativity, defined as confirmed ≥ 1 log10 between two consecutive positive samples in a patient who was previously tested as MRD negative
  * Death

SECONDARY OUTCOMES:
Tolerability of treatment | from FPFV until LPLV [4 years]
  cumulative occurence of CTCAE grade 3 and grade 4 adverse events
Remission (CR/CRi/CRh) rate | from FPFV until LPLV [4 years]
  CR/CRi/CRh rate is defined as the proportion of patients, who achieved a CR or CRi or CRh during study participation.
molecular response rate | from FPFV until LPLV [4 years]
  Proportion of patients with absence of detectable NPM1 mutant transcripts or with detectable NPM1 mutant transcripts who do not meet any of the definitions of molceular failure during study participation.
molecular persistence rate | from FPFV until LPLV [4 years]
  Proportion of patients with detectable NPM1 mutant transcripts present after four cycles of treatment with less than a 4 log10 reduction from baseline.
Rate of CR/CRi/CRh with MRD negativity | from FPFV until LPLV [4 years]
  Proportion of patients, who achieved a CR or CRi or CRh with NPM1-mutant transcripts/ABL1 transcripts <0.01% during study participation.
early mortality | from FPFV until LPLV [4 years]
  Early mortality is defined as death from any reason within 14, 30 and 60 days from day 1 of induction treatment.
Relapse-free survival (RFS) | from FPFV until LPLV [4 years]
  Relapse-free survival is defined as the time interval from date of first CR/CRi/CRh until either morphologic or molecular relapse or death in remission.
Overall survival (OS) | from FPFV until LPLV [4 years]
  Overall survival is defined as time interval from date of randomization until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Röllig, Prof., Principal Investigator — Technische Universität Dresden, Medical Faculty Carl Gustav Carus
Locations (18):
- Germany (18):
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Aachen, Aachen
  - Universitätsklinikum Augsburg, Augsburg
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universiätsklinikum Köln, Cologne
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Johann Wolfgang Goethe-Universität, Frankfurt am Main
  - Universitätsklinikum Halle, Halle
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Mannheim gGmbH, Mannheim
  - Philipps-Universität Marburg Fachbereich Medizin, Marburg
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg-Nord, Nuremberg
  - Krankenhaus Barmherzige Brüder, Regensburg
  - Robert-Bosch-Krankenhaus, Stuttgart